CLINICAL TRIAL: NCT00063895
Title: A Pharmacogenetic and Pharmacodynamic Study of Erlotinib (OSI-774) Toxicity in Patients With Advanced Solid Tumors
Brief Title: Erlotinib in Treating Patients With Advanced Non-Small Cell Lung Cancer, Ovarian Cancer, or Squamous Cell Carcinoma of the Head and Neck
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-03097; 12202A; U01CA069852 (NIH); U01CA070095 (NIH)
Record Dates: First submitted 2003-07-08; First posted 2003-07-09 (Estimated); Last update posted 2013-01-09 (Estimated); Status verified 2013-01

CONDITIONS: Recurrent Non-small Cell Lung Cancer; Recurrent Ovarian Epithelial Cancer; Recurrent Squamous Cell Carcinoma of the Hypopharynx; Recurrent Squamous Cell Carcinoma of the Larynx; Recurrent Squamous Cell Carcinoma of the Lip and Oral Cavity; Recurrent Squamous Cell Carcinoma of the Nasopharynx; Recurrent Squamous Cell Carcinoma of the Oropharynx; Stage III Squamous Cell Carcinoma of the Hypopharynx; Stage III Squamous Cell Carcinoma of the Larynx; Stage III Squamous Cell Carcinoma of the Lip and Oral Cavity; Stage III Squamous Cell Carcinoma of the Nasopharynx; Stage III Squamous Cell Carcinoma of the Oropharynx; Stage IIIA Non-small Cell Lung Cancer; Stage IIIA Ovarian Epithelial Cancer; Stage IIIB Non-small Cell Lung Cancer; Stage IIIB Ovarian Epithelial Cancer; Stage IIIC Ovarian Epithelial Cancer; Stage IV Non-small Cell Lung Cancer; Stage IV Ovarian Epithelial Cancer; Stage IV Squamous Cell Carcinoma of the Hypopharynx; Stage IV Squamous Cell Carcinoma of the Nasopharynx; Stage IVA Squamous Cell Carcinoma of the Larynx; Stage IVA Squamous Cell Carcinoma of the Lip and Oral Cavity; Stage IVA Squamous Cell Carcinoma of the Oropharynx; Stage IVB Squamous Cell Carcinoma of the Larynx; Stage IVB Squamous Cell Carcinoma of the Lip and Oral Cavity; Stage IVB Squamous Cell Carcinoma of the Oropharynx; Stage IVC Squamous Cell Carcinoma of the Larynx; Stage IVC Squamous Cell Carcinoma of the Lip and Oral Cavity; Stage IVC Squamous Cell Carcinoma of the Oropharynx
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Carcinoma, Ovarian Epithelial; Squamous Cell Carcinoma of Head and Neck | interventions — Erlotinib Hydrochloride; Pharmacogenomic Testing

ARMS (1):
- Treatment (erlotinib hydrochloride) (Experimental): Patients receive oral erlotinib on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: erlotinib hydrochloride; Other: pharmacological study; Other: pharmacogenomic studies; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: erlotinib hydrochloride — Given PO
  Other Names: CP-358,774; erlotinib; OSI-774
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies
Other: pharmacogenomic studies — Correlative studies
  Other Names: Pharmacogenomic Study
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase I/II trial is studying the side effects of erlotinib and to see how well it works in treating patients with metastatic or unresectable non-small cell lung cancer, ovarian cancer, or squamous cell carcinoma (cancer) of the head and neck. Erlotinib may stop the growth of tumor cells by blocking the enzymes necessary for their growth

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine if a significant correlation exists between the length of the CA dinucleotide repeat polymorphism in the EGFR gene and observed toxicity in patients treated with OSI-774.

SECONDARY OBJECTIVES:

I. To study the pharmacodynamic effects of OSI-774 on EGFR activity and MAP kinase signaling using skin as a surrogate tissue.

II. To determine if interindividual variation of OSI-774 pharmacokinetics is related to a previously described CYP3A5 genetic polymorphism.

III. To evaluate whether toxicity or inhibition of EGFR phosphorylation correlates with OSI-774 AUC in patients treated with OSI-774.

IV. To describe the observed anti-tumor response and toxicities in patients with advanced solid tumors treated with single agent fixed dose of OSI-774.

OUTLINE: This is a multicenter study. Patients are stratified according to length of CA dinucleotide repeat polymorphism (short vs medium vs long).

Patients receive oral erlotinib on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed metastatic or unresectable non-small cell lung cancer, squamous cell carcinoma of the head and neck, or ovarian cancer
* Eligible patients must have been off previous anticancer therapy including chemotherapy, radiotherapy, biological therapy, or other investigational therapy for at least 4 weeks before study entry (6 weeks if prior therapy included nitrosoureas or mitomycin C)
* ECOG performance status =< 2 (Karnofsky >= 60%)
* Life expectancy of greater than 12 weeks
* Leukocytes >= 3,000/ul
* Absolute neutrophil count >= 1,500/ul
* Platelets >= 100,000/ul
* Total bilirubin within normal institutional limits
* Creatinine within normal institutional limits OR creatinine clearance > 60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal
* Patients must have measurable or assessable disease
* The effects of OSI-774 on the developing human fetus are unknown; for this reason women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier; patients with prior treatment with small molecule inhibitors of EGFR, including erlotinib and gefitinib, are not eligible for this study
* Patients may not be receiving any other investigational agents
* Patients with uncontrolled brain metastasis; patients with brain metastases must have stable neurologic status following local therapy (surgery or radiation) for at least 4 weeks, and must be without neurologic dysfunction that would confound the evaluation of neurologic and other adverse events
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to OSI-774
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study because OSI-774 is an agent with the potential for teratogenic or abortifacient effects; because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with OSI-774, breastfeeding should be discontinued if the mother is treated with either agent
* HIV-positive patients receiving combination anti-retroviral therapy are excluded from the study because of possible pharmacokinetic interactions with OSI-774 or other agents administered during the study; appropriate studies will be undertaken in patients receiving combination anti-retroviral therapy when indicated
* Patients with significant ophthalmologic abnormalities, including: severe dry eye syndrome, kerato-conjunctivitis sicca, Sjogren's syndrome, severe exposure keratopathy, disorders that might increase the risk for epithelium-related complications (e.g. bullous keratopathy, aniridia, severe chemical burns, neutrophilic keratitis); patients with mild forms of any of the above, an asymptomatic history, or a normal ophthalmologic examination may be considered for inclusion at the discretion of the investigator; an ophthalmologic exam is not needed prior to this study unless clinically indicated; patients with treatable conditions (e.g. infectious keratitis/conjunctivitis, allergic conjunctivitis) may be reevaluated for study eligibility after treatment or resolution of the condition; use of contact lenses during the course of this trial may increase the risk of corneal complications and will be strongly discouraged
* Serious, non-healing wound ulcer, or bone fracture
* Major surgical procedure, open biopsy or significant traumatic injury within 14 days prior to Day 1; following such procedures or injuries, wound healing should be evident prior to initiation of therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2003-04; Primary Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
Rate of diarrhea and skin rash across the short, medium, and long genotype frequencies of the CA polymorphism | Baseline
  Compared using Armitage's test for a trend in proportions. In the event that the relationship between toxicity and length of the polymorphism is not monotone, a two degree-of-freedom chisquare test will be used in place of the trend test. The number of CA repeats treated as a continuous variable by averaging the number of repeats on each chromosome. Logistic regression analysis will then be performed to model the probability of toxicity as a function of the average length.
Rate of diarrhea and skin rash across the short, medium, and long genotype frequencies of the CA polymorphism | Week 6
  Compared using Armitage's test for a trend in proportions. In the event that the relationship between toxicity and length of the polymorphism is not monotone, a two degree-of-freedom chisquare test will be used in place of the trend test. The number of CA repeats treated as a continuous variable by averaging the number of repeats on each chromosome. Logistic regression analysis will then be performed to model the probability of toxicity as a function of the average length.

SECONDARY OUTCOMES:
Pharmacodynamic effects of erlotinib hydrochloride on EGFR activity and MAP kinase signaling | Week 1
Observed anti-tumor responses | Up to 4 years
  Number of patients with complete or partial tumor responses and will be tabulated; 95% confidence intervals will be generated.
All observed toxicities | Up to 4 years
  The frequency of adverse events will be tabulated; 95% confidence intervals will be generated.
Erlotinib hydrochloride AUC | Baseline, 0.5, 1, 2, 4, and 6 h after initiation, and pre-treatment days 15 and 29
  Compared with incidence of toxicity in patients with at least one 3A5*1 allele to those with no 3A5*1 allele using two-sample t and chi square tests, respectively. The relationship between toxicity and AUC evaluated by fitting ordinal (proportional odds) logistic regression models in which the grade of toxicity is the dependent variable and AUC is the independent or predictor variable. If the proportional odds model does not provide a good fit to the data then the toxicity grade will be dichotomized and analyzed using and analyzed using ordinary logistic regression.

CONTACTS AND LOCATIONS:
Overall Officials: Charles Rudin, Principal Investigator — University of Chicago Comprehensive Cancer Center
Locations (1):
- University of Chicago Comprehensive Cancer Center, Chicago, Illinois, United States